CLINICAL TRIAL: NCT02851459
Title: Tailoring of Vaccine-Focused Messages: Moral Foundations and Disease Salience - Part 1
Brief Title: Tailoring of Vaccine-Focused Messages: Moral Foundations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Saad B. Omer, MBBS, MPH, PhD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00087211
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Childhood Vaccinations
Keywords: Vaccines
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Morally Congruent Message (Experimental): Participants randomized to this arm will receive a vaccine-related message developed to appeal to their three most-emphasized moral foundations.
  Interventions: Behavioral: Baseline Survey; Behavioral: Pre-intervention Survey; Behavioral: Morally Congruent Message; Behavioral: Post-Intervention Survey
- Morally Non-Congruent Message (Experimental): Participants randomized to this arm will receive a vaccine-related message developed to appeal to their three least-emphasized moral foundations.
  Interventions: Behavioral: Baseline Survey; Behavioral: Pre-intervention Survey; Behavioral: Morally Non-Congruent Message; Behavioral: Post-Intervention Survey
- Control Message (Sham Comparator): Participants randomized to the control arm will be provided with a short passage about the costs and benefits of bird feeding.
  Interventions: Behavioral: Baseline Survey; Behavioral: Pre-intervention Survey; Behavioral: Control Message; Behavioral: Post-Intervention Survey

INTERVENTIONS:
Behavioral: Baseline Survey — The baseline survey contains questions regarding level of existing vaccine hesitancy (Parent Attitudes about Childhood Vaccines (PACV) short scale and HealthStyles questions), demographic information, and intent to vaccinate their children. All study surveys will be completed on an electronic device.
Behavioral: Pre-intervention Survey — Participants will be contacted two weeks after completing the baseline survey to answer questions about their moral beliefs. The survey will include questions form the Moral Foundations Questionnaire as well as additional questions. An algorithm will calculate the participant's moral matrix based on answers to these questions.
Behavioral: Morally Congruent Message — Intervention messages consist of four short paragraphs. The first three focus on how getting vaccinated helps uphold specific moral foundations. The fourth summarizes the contents of the prior paragraphs.
  Participants randomized to the morally congruent arm will receive a vaccine-related message developed to appeal to their three most-emphasized moral foundations. The first paragraph focuses on the most emphasized foundation, the second on the third-most emphasized, and the third on the second-most emphasized.
  Other Names: Morally Congruent Vaccine Focused Message
  Arms: Morally Congruent Message
Behavioral: Morally Non-Congruent Message — Intervention messages consist of four short paragraphs. The first three focus on how getting vaccinated helps uphold specific moral foundations.
  Participants randomized to the morally non-congruent arm will receive a vaccine-related message developed to appeal to their three least-emphasized moral foundations. The first paragraph focuses on the least emphasized foundation, the second on the third-least emphasized, and the third on the second-least emphasized.
  Other Names: Morally Non-Congruent Vaccine Focused Message
  Arms: Morally Non-Congruent Message
Behavioral: Control Message — Participants randomized to the control arm will be provided with a short passage about the costs and benefits of bird feeding.
  Arms: Control Message
Behavioral: Post-Intervention Survey — Immediately after reading the randomly assigned message participants will complete a follow-up survey assessing level of existing vaccine hesitancy (PACV short scale and HealthStyles questions) and intent to vaccinate their children.

SUMMARY:
This study is the first phase of a trial examining decision making about vaccines. This phase tests the impact of targeted vaccine-focused health messages on vaccine beliefs held by parents of young children and pre-adolescents. The participant's vaccine beliefs will be assessed at baseline. Two weeks later, the participant's moral matrix will be assessed. A vaccine-related message that appeals to the individual's three most or least emphasized moral foundations will then be presented. Immediately afterwards, vaccine beliefs will be assessed to determine the impact of the message.

DETAILED DESCRIPTION:
Vaccination of young children helps protect this population against a variety of diseases. Children are especially at risk for contraction of and complications from diseases due to their vulnerable immune systems. New evidence-based messages are needed to maintain and increase vaccination uptake among this group. An emphasis on different values is related to decisions parents make about vaccines. The purpose of this study is to develop, implement, and evaluate messages that focus on different aspects of values to impact vaccination attitudes among parents of young children.

Parents emphasize different moral foundations when deciding whether or not to vaccinate children. Based on this research, a messaging intervention with parents of children who are 12 years of age or younger will be conducted. These messages will aid in assessment of how different moral foundations impact attitudes towards vaccination and intent to vaccinate.

This study tests the impact of targeted vaccine-focused health messages on vaccine beliefs held by parents of young children and pre-adolescents. The participant's vaccine beliefs will be assessed at baseline. Two weeks later, the participant's moral matrix will be assessed. A vaccine-related message that appeals to the individual's three most or least emphasized moral foundations will then be presented. Immediately afterwards, vaccine beliefs will be assessed to determine the impact of the message.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one child ≤ 12 years of age
* Reside in the United States

Exclusion Criteria:

* Have previously participated in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 850 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Overall change in attitude towards vaccines | Week 2
  Number of caregivers experiencing a change in attitude towards vaccines.
Intent to have their children vaccinated | Week 2
  Number of caregivers opting to have their children vaccinated.

CONTACTS AND LOCATIONS:
Overall Officials: Saad B Omer, BBS, MPH, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University School Of Public Health - Only Online Recruitment, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No